CLINICAL TRIAL: NCT01213940
Title: Vascular Endothelium Changes After Bariatric Surgery
Brief Title: Vascular Endothelium Changes After Bariatric Surgery (Endothelial Progenitor Cells)
Acronym: EPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Alabama (Other)
Collaborators: American Society for Metabolic and Bariatric Surgery (Other)
Responsible Party: Principal Investigator, William Richards, Professor and Chairman of the Department of Surgery, University of South Alabama
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10-131
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Weight Reduction Programs; Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- baratric surgery (Other): surgery vs.weight loss program 6 months prior to bariatric surgery
  Interventions: Procedure: bariatric surgery
- pre-bariatric weight loss program (Other): weight loss program prior to bariatric surgery
  Interventions: Behavioral: pre-bariatric weight loss program

INTERVENTIONS:
Behavioral: pre-bariatric weight loss program — standard 6 month physician directed pre-bariatric weight loss program
  Other Names: weight loss program
  Arms: pre-bariatric weight loss program
Procedure: bariatric surgery — bariatric surgery for weight loss
  Arms: baratric surgery

SUMMARY:
Improvement in cardiovascular mortality is related to changes in pathologic autoantibodies and in the number of circulating functional replicative competent endothelial progenitor cells (EPC's) after bariatric surgery.

DETAILED DESCRIPTION:
Same as above

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes, Glucose > 200mg/dl, currently be ing treated with oral medications and HGA1c . 6.5, and BMI .35.

Exclusion Criteria:

* Type 1 Diabetes

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William O Richards, MD, Principal Investigator — University of South Alabama, Department of Surgery
Locations (1):
- University of South Alabama, Mobile, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Baratric Surgery | Pre-bariatric Weight Loss Program
Started | 14 | 6
Completed | 14 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Baratric Surgery | Pre-bariatric Weight Loss Program | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 2 | 2 | 4
body mass index [Mean (Full Range); unit: kg/m2] | 46.6 [39.4 to 69.4] | 44.1 [38.4 to 73.3] | 45.9 [38.4 to 73.3]

OUTCOME MEASURES:

1. Primary Outcome: Change in Late Outgrowth Endothelial Progenitor Colonies
Description: Primary outcome is the change in Late outgrowth endothelial progenitor colonies 12 months after enrollment to surgery (LRYGB) or to standard medical therapy (SMT).
Time Frame: 24 months
Population: Study population of patients undergoing bariatric surgery compared to a group of morbidly obese patients undergoing medical diet therapy pre bariatric surgery
Measure: Mean (Standard Error); unit: LOEPC colonies
Groups:
- Bariatric Surgery: surgery vs, weight loss program 6 months prior to bariatric surgery
Arm/Group | Bariatric Surgery | Pre-bariatric Weight Loss Program
Number analyzed (Participants) | 14 | 6
LOEPC colonies
  LOEPC Colonies baseline | 0.3 (0.1) | 0.2 (0.1)
  LOEPC colonies 24 months post bariatric surgery | 3.1 (.9) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Bariatric Surgery vs Pre-bariatric Weight Loss Program; one -way ANOVA was used for the analysis; Test type: Equivalence — 95% confidence limit from standard deviation of mean; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: baseline to 6 months
Description: Serious adverse events were identified through regular investigator assessment.
Arm/Group | Baratric Surgery | Pre-bariatric Weight Loss Program
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6
Other Adverse Events (participants affected / at risk) | 0/14 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No